CLINICAL TRIAL: NCT02351011
Title: Human Autologous Mesenchymal Stromal Cells for the Treatment of Mid to Late Stage Knee Osteoarthritis
Brief Title: Human Autologous MSCs for the Treatment of Mid to Late Stage Knee OA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jas Chahal (Other)
Responsible Party: Sponsor-Investigator, Jas Chahal, Orthopaedic Surgeon, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MSC-001
Record Dates: First submitted 2015-01-20; First posted 2015-01-30 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): 1 x 10^6 MSCs
  Interventions: Biological: 1 x 10^6 MSCs
- Cohort 2 (Experimental): 10 x 10^6 MSCs
  Interventions: Biological: 10 x 10^6 MSCs
- Cohort 3 (Experimental): 50 x 10^6 MSCs
  Interventions: Biological: 50 x 10^6 MSCs

INTERVENTIONS:
Biological: 1 x 10^6 MSCs — Autologous, bone-marrow derived MSCs
  Other Names: Mesenchymal Stromal Cells (MSCs)
  Arms: Cohort 1
Biological: 10 x 10^6 MSCs — Autologous, bone-marrow derived MSCs
  Other Names: Mesenchymal Stromal Cells (MSCs)
  Arms: Cohort 2
Biological: 50 x 10^6 MSCs — Autologous, bone-marrow derived MSCs
  Other Names: Mesenchymal Stromal Cells (MSCs)
  Arms: Cohort 3

SUMMARY:
Osteoarthritis (OA) is one of the most common forms of arthritis. It is a lasting condition in which the material that cushions the joints, called cartilage, breaks down. This causes the bones to rub against each other, causing inflammation, stiffness, pain and loss of joint movement. Currently, there are few effective treatments available for patients suffering from OA.

Mesenchymal stem cells (MSCs) are cells that have the ability to self-regenerate, which means they have the ability to make copies of themselves and to turn into other kinds of cells (e.g. cartilage cells). Stem cell science shows much promise for the future treatment of osteoarthritis, but much of the research is still in the early stages. In this study, researchers want to determine the safety of MSCs that a patient can tolerate without causing side effects. This will be done by starting at a low dose of MSCs and moving on to the next higher dose level provided there are no safety concerns. Researchers will also be looking at the function of the knee over time, which may give them some insight on the usefulness of MSCs as a treatment option.

DETAILED DESCRIPTION:
The trial is a non-randomized, open-label, dose escalation phase I/II clinical trial. A total of 12 participants will be enrolled - patients will be treated in cohorts of 3 to determine the safety and preliminary efficacy of autologous, ex-vivo expanded bone-marrow derived MSC injected into the knee joint in patients with moderate to advanced knee osteoarthritis.

A minimum of three evaluable patients will be entered at each dose level until the maximum tolerated dose (MTD) is reached. Toxicity will be evaluated and graded according to the Common Terminology Criteria (CTC) for Adverse Events, as Grade 3-4. If a patient is discontinued due to a grade 3 or 4 adverse event (i.e. dose-limiting toxicity, DLT), an additional patient will be enrolled at the same dose level to ensure that a minimum of 3 patients are evaluated. If 0/3 patients experience dose-limiting (DLT) at a given dose level, then the dose will be escalated for next cohort of 3 patients. If 1/3 patients experience DLT at a given dose level, then an additional 3 patients will be treated at that dose level. If no other patient experiences a DLT, dose escalation will continue. If DLT occurs in 2/3 or 2/6 patients, dose escalation will stop and the prior dose level will be declared the MTD for the MSC cell infusions in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 40-65 years of age with symptomatic moderate to severe (Kellgren-Lawrence III or IV) primary osteoarthritis of the knee
2. Failed conservative management including physical therapy, bracing and/or oral anti-inflammatories for a minimum of six months
3. No history of prior intra-articular cortisone, hyaluronic acid, or platelet-rich plasma injection within the previous six months
4. No history of prior arthroscopic knee surgery or open knee surgery on the ipsilateral side within the past year
5. Adequate bone marrow, liver, and renal functions
6. Body weight >40 kg
7. Body Mass Index <30
8. Negative for (HIV, HTLV1&2, Hep A, B, C, syphilis) infection as determined by approved serological testing
9. Negative for pregnancy as determined by a serum pregnancy test. Females of childbearing potential will be required to practice abstinence or use an effective form of contraception for 12 months following their MSC injection.
10. Fluid > 1 cm within the lateral recess of the suprapatellar pouch at the level of the superior pole of the patella with the knee extended.

Exclusion Criteria:

1. Patients with clinically unstable knee due to the presence of a complete anterior cruciate ligament, posterior cruciate ligament, medial collateral ligament and/or posterolateral corner tear
2. Patients with varus or valgus malalignment >5 degrees as measured by 4 foot standing antero-posterior radiographs
3. Patients with a history of a previous subtotal medial or lateral meniscectomy
4. Patients with a history of septic arthritis in the affected joint
5. Patients with a history of a prior intra-articular knee fracture
6. Severe bleeding diathesis
7. Contraindication to bone marrow aspiration and/or biopsy
8. Active infection
9. Bone marrow failure
10. Cytopenia
11. Patients who have previously received radiotherapy to the pelvis
12. Patients who have been on chemotherapy from within a year of the date of informed
13. Patients with positive serological test for (HIV, HTLV1&2, Hep A, B, C, syphilis)
14. Pregnancy or risk of pregnancy (this includes participants that are not willing to practice active contraception for the duration of the study)
15. Patients with unforeseen conditions that are deemed unsafe or inappropriate for the study (e.g. patients who are claustrophobic and cannot undergo an MRI) as per the discretion of the principal investigator

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Safety as determined by the occurrence of local and systemic adverse events and/or serious adverse events. | 1 to 5 years
  Safety as determined by the occurrence of local and systemic adverse events and/or serious adverse events.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 1 year
  Knee-joint specific function
Marx Activity Scale (Patient-reported activity) | 1 year
  Patient-reported activity
Short-Form 36 (Health-related quality of life) | 1 year
  Health-related quality of life
Whole Organ MRI Score (WORMS), Gadolinium-enhanced MRI, T2 Mapping (To assess joint structure, inflammation, and cartilage status over time) | 1 year
  To assess joint structure, inflammation, and cartilage status over time
Cartilage oligomeric matrix protein (COMP) | 1 year
  Serum marker of cartilage metabolism
Hyaluronic acid (HA) | 1 year
  Serum pro-inflammatory marker
C-terminal telopeptide of type II collagen (CTXII) | 1 year
  Urine marker of cartilage metabolism
Types I and II collagen cleavage (C1,2C) | 1 year
  Urine marker of cartilage metabolism
Type II collagen cleavage (C2C) | 1 year
  Urine marker of cartilage metabolism
IL-6/TNFα/IL-15 | 1 year
  Synovial fluid pro-inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Jas Chahal, MD, MSc, Principal Investigator — Arthritis Program, Toronto Western Hospital; Sowmya Viswanathan, PhD, Principal Investigator — Arthritis Program, Toronto Western Hospital & Philip S. Orsino Facility for Cell Therapy
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada